CLINICAL TRIAL: NCT05318950
Title: A nUtrition and Lifestyle Intervention in Patients With Pulmonary Arterial HypertensIon: Effect on quaLity of Life
Brief Title: A nUtrition and Lifestyle Intervention in Patients With Pulmonary Arterial HypertensIon
Acronym: UPHILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Reinier de Graaf Groep (Other); Janssen-Cilag B.V. (Industry)
Responsible Party: Principal Investigator, A. Vonk Noordegraaf, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NL66484.029.18
Record Dates: First submitted 2021-12-10; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Nutrition; Lifestyle
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomisation control and E-learning Randomisation Diet A and B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention
- E-learning (Experimental): E-learning: 8 lessons about nutrition and lifestyle
  Interventions: Behavioral: E-learning
- Diet A (Experimental): MedDASH diet (55% carbohydrates, 25% amino acids, 20% fatty acids)
  Interventions: Behavioral: E-learning; Dietary Supplement: Diet
- Diet B (Experimental): MedDASHfat diet (10% carbohydrates, 25% amino acids, 65% fatty acids)
  Interventions: Behavioral: E-learning; Dietary Supplement: Diet

INTERVENTIONS:
Behavioral: E-learning — 8 lessons about nutrition and lifestyle
  Arms: Diet A; Diet B; E-learning
Dietary Supplement: Diet — Diet A: MedDASH diet (55% carbohydrates, 25% amino acids, 20% fatty acids) Diet B: MedDASHfat diet (10% carbohydrates, 25% amino acids, 65% fatty acids)
  Arms: Diet A; Diet B

SUMMARY:
Rationale: Nutrition and lifestyle interventions are currently not implemented in usual clinical care of PAH-patients. Mainly because there is little known on the relation between pathology, nutrition and lifestyle. Patients who suffer from Pulmonary Arterial Hypertension feel insecure about their nutrition and lifestyle. The investigators hypothesize that an intervention on nutrition and lifestyle can improve the patients' quality of life.

Objective: To explore the effect of a nutrition and lifestyle intervention on quality of life for patients suffering from PAH.

Study design: Investigator initiated intervention study with control group. Study population: investigators aim to include 70 patients (18 - 80 years) with idiopathic, hereditable or drug related PAH, who have been stable for at least three months and are self-sufficient and/or have a family who's willing to participate in the lifestyle changes.

Intervention (if applicable): Nutritional status, - education, - intervention and - compliance.

Main study parameters/endpoints: This is an intervention study in which the investigators will asses the effect of a nutrition and lifestyle intervention on quality of life measured by SF-36 overall outcome with a significant difference of 6.35.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden for the patient exists of 12 extra visits to the hospital and contact moments, over a period of 11 months, as well compliance to the diet and lifestyle. There is minimal risk in participation.

DETAILED DESCRIPTION:
Baseline nutritional assessment

Nutritional education:

8 online lessons containing information about nutrition, lifestyle and general health with complementary tips regarding PH. All participants recieve workbook with assignments.

Nutritional intervention:

Group A: MedDASH diet (55% carbohydrates, 25% amino acids, 20% fatty acids) Group B: MedDASHfat diet (10% carbohydrates, 25% amino acids, 65% fatty acids) Control group: no diet.

Follow-up:

Patients in intervention arm followed for a period of 6 months to assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PAH, hereditable PAH or drug related PAH
* Age between 18 and 80
* NYHA II or III and stable for at least 3 months, determined by a stable 6minute walk test with a difference of <10%.
* Self-sufficient and/or compliance from partner and/or family
* Creatinine > 30 ml/min
* Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria:

* - Pregnant subjects
* Fat percentage < 10% > 50 %
* One or more of the following comorbidities: diabetes mellitus type one or two, clinically relevant thyroid disease
* Known history of noncompliance considering therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline (week 0), after nutritional education (week 10), after nutritional intervention (week 24), after follow up (week 48)
  To asses quality of life, the SF-36 questionnaire is used.

SECONDARY OUTCOMES:
Change in nutritional intake | Baseline (week 0), after nutritional education (week 10), after nutritional intervention (week 24), after follow up (week 48)
  To asses dietary intake a food frequency questionnaire is used (HELIUS)
Change in vitamin and mineral status | Baseline (week 0), after nutritional education (week 10), after nutritional intervention (week 24), after follow up (week 48)
  A complete serum analyses is performed to asses vitamin and mineral status.

OTHER OUTCOMES:
Change in exercise capacity | Baseline (week 0), after nutritional intervention (week 24), after follow up (week 48). The Fitbit is worn by intervention group over total study time (48 weeks)
  To determine exercise capacity subjects have to perform a six minute walking test
Change in heart rate variability | Baseline (week 0), after nutritional intervention (week 24), after follow up (week 48). The Fitbit is worn by intervention group over total study time (48 weeks)
  To determine heart rate variability all patients will receive a Fitbit smartwatch.
Change in daily activity | Baseline (week 0), after nutritional intervention (week 24), after follow up (week 48). The Fitbit is worn by intervention group over total study time (48 weeks)
  To determine changes in daily activity the number of steps will be assess by a Fitbit smartwatch

CONTACTS AND LOCATIONS:
Overall Officials: Anton Vonk Noordegraaf, prof. dr., Principal Investigator — VUMC
Locations (1):
- VU medical center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data of the study will be kept by the principal investigators and will be available for regulatory authorities. Subjects' personal data will be stored confidentially according to institutional routine. In principle, results will be published in peer-reviewed international journals.